CLINICAL TRIAL: NCT06844604
Title: Life Cylce Assessment (LCA) for Different Minimal Invasive Surgical Techniques: A Comparison of Robotic vs . Laparoscopic vs Open Colorectal Operation and Identification of Most Effective Carbon Foot Print Reduction Targets.
Brief Title: Carbon Footprint Assessment for Robotic, Laparoscopic and Open Colorectal Operations to Enhance Environmental Sustainability
Acronym: CARE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CARE25
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Operations
Keywords: colorectal operations; CO2 footprint; LCA; robotic colorectal surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- robotic colorectal procedures
  Interventions: Procedure: robotic colorectal procedures
- laparoscopic colorectal procedures
  Interventions: Procedure: laparoscopic colorectal procedures
- open colorectal procedures
  Interventions: Procedure: open colorectal procedures

INTERVENTIONS:
Procedure: robotic colorectal procedures — any colorectal procedure planed robot-assisted
  Groups: robotic colorectal procedures
Procedure: laparoscopic colorectal procedures — any colorectal procedure planed laparoscopically
  Groups: laparoscopic colorectal procedures
Procedure: open colorectal procedures — any colorectal procedure planed open
  Groups: open colorectal procedures

SUMMARY:
The goal of this study is to conduct a life cycle assessment of robotic, laparoscopic and open colorectal procedures and compare their climate impact. Further the investigators want to identify major targets for possible reduction in the CO2 footprint in colorectal procedures. The main questions are:

Researchers will identify used and prepared materials and instruments for the individual procedures and weigh them individually. SimaPro databases will help calculate the carbon footprints for the used instruments. Additionally, energy waste will be measured and carbon footprint of anesthesia will be estimated with previous existing data from other studies.

DETAILED DESCRIPTION:
Background Effective reduction of greenhouse gas (GHG) emissions as the key driver for climate change has to be the primary target of sustainable economics in the 21st century . The carbon footprint is calculated by the direct and indirect attributable GHGs emitted during a process, production cycle, or from an institution, such as a hospital.[1] The main metric for calculating the carbon footprint is the CO2 equivalent (CO2eq). In Switzerland, about 6-7% of all CO2 emissions come from the healthcare system. Most CO2 emissions come from hospitals, followed by medical treatments.

A large contributor to hospitals' carbon footprints are operating rooms. The high energy demand, anesthetics, and the production of single-use devices and instruments are significant climate-related hotspots in the operating field. However, the life cycle assessment (LCA) varies considerably based on factors such as the type and modality of the operation, among other variables. To date, only a few direct comparisons of the climate impact between surgical modalities, such as open, laparoscopic, and robot-assisted procedures, have been studied.

In this study, the investigators aim to compare the three modalities of visceral operations and their impact on the carbon footprint. As previously mentioned, a major component of the high GHG production in operating rooms is the high energy demand and needed resources. The best method to calculate the climate impact is the use of LCA.

Within an LCA, climate-related hotspots can be identified for each operation analyzed, which can provide possible ideas to reduce the carbon footprint of operating rooms and their impact on climate change.

Methods For this comparison, the investigators will conduct an LCA for each operation observed and compare it among the three different modalities: robotic, laparoscopic and open colorectal procedures.

The LCA includes direct and indirect GHG emissions throughout a product's lifetime, as well as energy consumption during the operation. This encompasses the raw materials used, emissions during production and transportation, and the accumulated waste. A life cycle inventory (LCI) collects LCAs for all instruments and products used during the procedure and during preparation.

Used surgical instruments, drapes, gloves and gowns will be registered in the prefabricated datasheet during the observed colorectal operation. Single-use equipment recorded in the datasheet will be weighed individually before usage. During the procedure the investigators will then identify not used and used materials and instruments. Their packaging will be weighed after the operation to differentiate between packaging and absolute weight of used instrument. Using the manufacturer's information about raw material usage in each product, the investigators will calculate the CO2 footprint of the individual instruments and materials. In the Ecoinvent database with recorded CO2 emissions per kilogram of raw material will provide the necessary information to conduct LCAs for each product used in the operating room. This study will include sterile as well as non-sterile equipment used during preparing and performing the procedure. For reusable instruments, the investigators will estimate the total CO2 footprint, including the sterilization process, using average values from previous studies. Reusable instruments used for robotic operations is estimated to have a life span of around 10 to 15 sterilization processes. The estimated life cycle for laparoscopic reusable instruments is set to be around 100 sterilization processes. Other reusable surgical instruments that are commonly used are estimated to live up to 1000 sterilization cycles.

During the procedures the investigators will identify the majority of not used but prepared instruments. Additionally to the materials and instruments the investigators will record the used anesthetics for general anesthesia and with previous study calculate the estimated climate impact For the secondary research question the investigators will differentiate between used, opened and prepared equipment in the operating room during the procedure. The research team will therefore additionally identify material and instruments that were unpacked but not used during the procedures It is important to state, that only used and opened instruments and materials will be included in the calculation of the CO2 footprint.

To calculate the energy used during the operations, the kilowatt hours (kWh) needed during the procedure itself will be extracted as average energy consumption in the operating room where the surgery took place. The investigators will then calculate the CO2 footprint using information about the clinic's energy mix. Additionally, the research team will use standardized calculations for the CO2 footprint of anesthesia and hospital stay to estimate the value for the observed operations.

The raw data will be collected in an REDCAP database and further analyzed with the software SimaPro or OpenLCA. The investigators then estimate the related CO2 footprint per procedure. The mean CO2 footprint will afterwards be used to compare the three modality. For comparisons between groups, the research team will use the Mann-Whitney U test in R and RStudio. Climate impact will be estimated using the ReCiPe method.

Target The aim of the LCA robotic operation study is to compare the carbon footprint between robotic, laparoscopic and open colorectal procedures and to identify major targets for the reduction of CO2 emissions.

ELIGIBILITY:
Inclusion Criteria:

* Elective operations which are routinely performed robot-assisted, laparoscopic and open:

  * Only Colorectal procedures involving a bowel resection will be included (colectomies (right/left), anterior resections)
* General anesthesia
* Aged > 18 years
* ASA classification from I to III

Exclusion Criteria:

* Procedures, which were uncompleted due to complications
* Procedures, which switched modality (laparoscopic to open, robot-assisted to open)
* Emergency procedures (mainly laparoscopic, unforeseen risk factors that lead to a change of modality, higher volume of used compressions and other materials).
* Aged younger than 18
* ASA classification > III
* Vulnerable patient groups (pregnancy, patients with mental disability)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from primary care units that are in need of a colorectal surgery and fulfil the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of climate impact between robotic, laparoscopic and open colorectal procedures | 9 monts
  Conduct an analysis of the climate impact of the three modalities of modern visceral operation and the standardized hospital days after the observed surgeries using LCA and the ReCiPe method. Compare the three modalities.

SECONDARY OUTCOMES:
Identify major targets for possible reduction in the CO2 footprint in visceral procedures. | 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Clarunis, Basel
  - University Hospital of Basel, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huijbregts Mark A.J., Steinmann Zoran J.N., Eishout Pieter M. F., Stam Gea, Verones Francesca, ReCiPe2016: a harmonised life cycle impact assessment method at midpoint and endpoint level, The international Journal of Life Cycle Assessment, 02.01.2017
- [Background] Misrai V, Rijo E, Cottenceau JB, Zorn KC, Enikeev D, Elterman D, Bhojani N, De La Taille A, Herrmann TRW, Robert G, Pradere B. A Standardized Method for Estimating the Carbon Footprint of Disposable Minimally Invasive Surgical Devices: Application in Transurethral Prostate Surgery. Ann Surg Open. 2021 Sep 7;2(3):e094. doi: 10.1097/AS9.0000000000000094. eCollection 2021 Sep. PMID 37635829
- [Background] Woods DL, McAndrew T, Nevadunsky N, Hou JY, Goldberg G, Yi-Shin Kuo D, Isani S. Carbon footprint of robotically-assisted laparoscopy, laparoscopy and laparotomy: a comparison. Int J Med Robot. 2015 Dec;11(4):406-12. doi: 10.1002/rcs.1640. Epub 2015 Feb 22. PMID 25708320
- [Background] Sapuan S.M., Ilyas R. A., Asyraf M. R. M., Carbon footprint in Healthcare, Springer, 2022
- [Background] Rodriguez-Jimenez L, Romero-Martin M, Spruell T, Steley Z, Gomez-Salgado J. The carbon footprint of healthcare settings: A systematic review. J Adv Nurs. 2023 Aug;79(8):2830-2844. doi: 10.1111/jan.15671. Epub 2023 May 17. PMID 37198974
- [Background] swissinfo.ch, health system causes too high CO2 emissions, says top Swiss doctor, SWI swissinfo.ch, 10.27.2023
- [Background] Wiedmann Thomas, Minx Jan, A definition of carbon footprint, Nova science Publishers, 2007
- See also: Related Info — https://www.swissinfo.ch/eng/business/health-system-causes-too-high-co2-emissions-says-top-swiss-doctor/48929594
- See also: Related Info — https://medizin.unibas.ch/en/default-pages/news/details/this-was-the-event-sustainability-in-the-healthcare-sector/
- See also: Related Info — https://www.iso.org/standard/37456.html